CLINICAL TRIAL: NCT01513057
Title: An Open-label, Balanced, Randomized, Two-treatment, Two-period, Two Sequence, Single Dose, Crossover, Bioequivalence Study in Healthy, Adult,Human, Male Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Mycophenolate Mofetil 250 mg Capsule, Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 466-08
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: bioequivalence; Mycophenolate Mofetil; crossover
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolate Mofetil (Experimental): Mycophenolate Mofetil 250 mg capsules of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Mycophenolate Mofetil
- Cellcept (Active Comparator): Cellcept 250 mg capsules of Roche Laboratories Inc.
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil 250 mg capsules of Dr. Reddy's Laboratories Limited
  Arms: Mycophenolate Mofetil
Drug: Mycophenolate Mofetil — 250 mg capsules of Roche Laboratories Inc.
  Other Names: Cellcept
  Arms: Cellcept

SUMMARY:
An open-label, balanced, randomized, two-treatment, two-period, two sequence, single dose, crossover, bioequivalence study of Mycophenolate mofetil 250 mg Capsule of Dr. Reddy's Laboratories limited, comparing with that of Cellcept 250 mg Capsule of Roche Laboratories in healthy, adult, human, male subjects under fed conditions.

DETAILED DESCRIPTION:
This was an open-label, balanced, randomized, two-treatment, two-sequence, two-period, single dose, crossover bioequivalence study in healthy, adult, human, male subjects under fed conditions.64 healthy male adults were enrolled.A washout period of 07 days was maintained between the successive dosing days.One capsule containing mycophenolate mofetil 250 mg was administered orally with 240 mL water in sitting posture, after an overnight fast of at least 10 hours in each period. This activity was followed by a mouth check to assess compliance to dosing. The subjects were not allowed to lie down for the first two hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, human male volunteers between 18 - 55 years of age (both inclusive) living in and around Ahmedabad city of western part of India.
* Having a Body Mass Index (BMI) between 18.5 - 24.9 (both inclusive), calculated as weight in kg/height in meter2.
* Have no significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12- lead ECG and X-ray chest recordings.
* Able to comply with the study procedures, in the opinion of the Principal investigator.
* Able to give voluntary written informed consent for participation in the study.

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to Mycophenolate mofetil or any related drug.
* Any disease or condition that compromised the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion of a medicine at any time with in 14 days before dosing in Period-I. In any such case subject selection was at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAID induced urticaria.
* A recent history of alcoholism (< 2 years) or of moderate (180 mL/day) alcohol use, or consumption of alcohol within 48 hours prior to receiving study medicine.
* Smokers, who smoked 10 or more than 10 cigarettes/day or inability to abstain from smoking during the study.
* Consumption of Grapefruits or its products within a period of 48 hours prior to dosing.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
* History of psychiatric disorders.
* A history of difficulty with donating blood.
* Donation of blood (1 unit or 350 mL) or receipt of an investigational product or participation in a drug research study within a period of 90 days prior to the first dose of study medicine. Elimination half-life of the study drug was taken into consideration for inclusion of the subject in the study.

Note: If subject had participated in a study in which blood loss was ≤ 200 mL, subject could be enrolled 60 days after the last sample of previous study.

* A positive hepatitis screen including hepatitis B surface antigen and HCV antibodies.
* A positive test result for HIV antibody and/or syphilis.
* An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medicine and throughout the subjects' participation in the study. In any such case subject selection was at the discretion of the Principal Investigator.

All the enrolled subjects satisfied all the above inclusion and exclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | pre-dose, 0.167, 0.333,. 0.500, 0.667, 0.833, 1.00, 1.25, 1.50, 1.75, 2.00, 2.25, 2.75, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, 60.00 and 72.00 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Kumar Jha, MD, Principal Investigator — Lambda Therapeutic Research Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, Gujarat, India